CLINICAL TRIAL: NCT03285984
Title: Plaque Removal Efficacy of Four Dentifrices in a Single Brushing Model
Brief Title: Ability of Four Toothpastes to Remove Plaque
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 202655
Record Dates: First submitted 2017-09-12; First posted 2017-09-18 (Actual); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque | interventions — Sodium Bicarbonate; Sodium Fluoride

STUDY DESIGN:
Intervention Model Description: The randomization schedule will indicate the treatment order sequence. Each subject will complete all four treatment regimens, one treatment regimen in each of the four treatment periods. This randomization will use a Williams Square layout and be provided by the Biostatistics Department, GSKCH.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test product 1 (Experimental): Participants will brush once (1.5g ± 0.05g of Test product 1), under supervision of study staff for one timed minute
  Interventions: Other: 67% Sodium Bicarbonate with 6 herbs plus 923parts per million (ppm) Sodium Fluoride
- Test product 2 (Experimental): Participants will brush once (1.5g ± 0.05g of Test product 2), under supervision of study staff for one timed minute
  Interventions: Other: 67% Sodium Bicarbonate without herbs plus 923 ppm Sodium Fluoride
- Test product 3 (Experimental): Participants will brush once (1.5g ± 0.05g of Test product 3), under supervision of study staff for one timed minute
  Interventions: Other: 62% Sodium Bicarbonate with 6 herbs and 5% w/w silica plus 923 ppm Sodium
- Test product 4 (Experimental): Participants will brush once (1.5g ± 0.05g of Test product 4), under supervision of study staff for one timed minute
  Interventions: Other: 0% Sodium Bicarbonate without herbs plus 923ppm Sodium Fluoride

INTERVENTIONS:
Other: 67% Sodium Bicarbonate with 6 herbs plus 923parts per million (ppm) Sodium Fluoride — Toothpaste containing 67 percent (%) Sodium Bicarbonate with 6 herbs plus 923parts per million (ppm) Sodium Fluoride
  Arms: Test product 1
Other: 67% Sodium Bicarbonate without herbs plus 923 ppm Sodium Fluoride — Toothpaste containing 67% Sodium Bicarbonate without herbs plus 923 ppm Sodium Fluoride
  Arms: Test product 2
Other: 62% Sodium Bicarbonate with 6 herbs and 5% w/w silica plus 923 ppm Sodium — Whitening Toothpaste containing 62% Sodium Bicarbonate with 6 herbs and 5% w/w silica plus 923 ppm Sodium
  Arms: Test product 3
Other: 0% Sodium Bicarbonate without herbs plus 923ppm Sodium Fluoride — Toothpaste containing 0% Sodium Bicarbonate without herbs plus 923ppm Sodium Fluoride
  Arms: Test product 4

SUMMARY:
The aim of this study is to evaluate and compare the plaque removal efficacy of four experimental toothpastes following a single timed brushing. Prior to each treatment visit, participants will abstain from oral hygiene for a period of 24 hours (+6hrs, -2hrs), immediately preceding a pre-brushing dental plaque evaluation. Participants will then brush once under supervision for one timed minute with each dentifrice after which re-disclosing and a post-brushing plaque assessment will be carried out.

DETAILED DESCRIPTION:
This study will be a single centre, randomized, controlled, examiner blind, four treatment, four period crossover design. At the screening visit, following provision of written informed consent, eligible participants will be provided with a washout toothpaste and toothbrush for use at home during the study and for at least 14 days prior to the first treatment visit.

Participants will then be scheduled to attend the first of four treatment visits a minimum of 14 days later. For each treatment visit, participants must abstain from oral hygiene for a period of 24 hours (+6hrs, -2hrs), immediately preceding the pre-brushing dental plaque evaluation. All the participants will undergo an oral soft tissue (OST) examination followed by disclosing and a dental plaque assessment.

At the treatment visit 1 pre-brushing plaque assessment, those who develop a sufficient amount of plaque (Turesky mean score ≥ 2.00) will be randomized to study treatment. Participants will then brush once (1.5 grams [g] ± 0.05g of assigned toothpaste), under supervision of study staff for one timed minute, with one of the four test toothpastes after which re-disclosing and a post-brushing plaque assessment will be carried out. Participants will be allowed to brush with the washout paste following the post assessment plaque assessments.

A minimum of three days washout period will follow each treatment period during which period Participants will brush with a commercial washout toothpaste. Participants will complete four treatment visits and will brush once with each of the four test toothpastes throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Aged at least 18 years
* Understands and is willing, able and likely to comply with all study procedures and restrictions
* Good general health with (in the opinion of the Investigator) no clinically significant and relevant abnormalities of medical history or dental history.
* Good dental health based on medical history and oral soft tissue examination at screening
* At least 20 gradable, natural, uncrowned teeth with both facial and lingual scoreable surfaces (gradable teeth are those where restorative materials cover less than 25% of the tooth surface graded)
* Plaque Score: Mean Turesky plaque score of ≥ 2.00 at treatment visit 1 pre-brushing plaque assessment

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study
* Women who are breast-feeding
* Antibiotic treatment within 14 days prior to Treatment Visit 1 or throughout the study
* Any other treatment that would interfere with the study results/conduct, at the discretion of the examiner or investigator
* Diabetes mellitus type I or II
* Any disease systemic or localized, dental or non dental, which could put the participant's health at risk or interfere with the study results/conduct, at the discretion of the examiner or investigator
* High levels of extrinsic stain or calculus deposits which might interfere with plaque assessments
* Dental condition/ disease requiring immediate treatment
* Pre-existing sensitivity to oral care products
* Severe gingivitis
* Periodontitis with pocket depth > 5mm affecting more than two teeth
* Moderate or severe recession
* Presence of orthodontic bands or appliances, extensive crowns, partial dentures, or fixed retainers on the maxillary or mandibular teeth
* Obvious active carious lesions needing immediate care
* Intra-oral decorative tattoos, or tongue and or lip piercing
* Oral lesions/manifestations that would impact on the outcome of the study
* Presence of oral or peri-oral ulceration including herpetic lesions at the time of screening or at baseline
* Known or suspected intolerance or hypersensitivity to the studymaterials (or closely related compounds) or any of their stated ingredients
* Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit
* Previous participation in this study
* Recent history (within the last year) of alcohol or other substance abuse
* Current use of Listerine or any antimicrobial mouth rinse containing Chlorhexidine or Cetrylpyridinium Chloride (CPC)
* Participant unwilling to abstain from using chewing tobacco (with or without tobacco)
* Participant unwilling to abstain from smoking on the morning prior to treatment visits
* An employee of the sponsor or the study site or members of their immediate family

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-03-27 (Actual); Primary Completion 2012-05-08 (Actual); Study Completion 2012-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Bosma ML, Milleman KR, Akwagyiram I, Targett D, Milleman JL. A randomised controlled trial to evaluate the plaque removal efficacy of sodium bicarbonate dentifrices in a single brushing clinical model. BDJ Open. 2018 Jun 4;4:17037. doi: 10.1038/s41405-018-0003-7. eCollection 2018. PMID 29971158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single center in the United States.
Pre-assignment Details: A Total of 56 participants were screened and randomized in the study. All 56 participants completed the study.
Groups:
- Overall Study: This was a single centre, randomized, controlled, examiner blind, four treatment, four period crossover design study. Each Participant received Test product 1 (Toothpaste containing 67 percent [%] sodium bicarbonate with 6 herbs plus 923 parts per million [ppm] sodium fluoride, Test product 2 (Toothpaste containing 67% sodium bicarbonate without herbs plus 923ppm sodium fluoride), Test product 3 (Whitening Toothpaste containing 62% Sodium Bicarbonate with 6 herbs and 5% weight by weight [w/w] silica plus 923ppm Sodium), and Test product 4 (Toothpaste containing 0% Sodium Bicarbonate without herbs plus 923ppm sodium fluoride).
Period: Overall Study
Arm/Group | Overall Study
Started | 56
Received Test Product 1 | 56
Received Test Product 2 | 56
Received Test Product 3 | 56
Received Test Product 4 | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants were included for baseline evaluation.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.1 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 51
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (Pre-brushing to Post-brushing) in Turesky Score After Single Supervised Use (Test Product 1 Versus [vs] Test Product 4) After 4 Weeks
Description: The dental examiner used Turesky Modification of the Quigley Hein Index to assess plaque on all gradable teeth.Overall plaque scores were calculated taking average over all tooth sites for participant.Plaque was first disclosed using dye solution followed by disclosing solution.They expectorated and rinsed with 10 milliliters (mL) water for 10 seconds (sec),expectorated again. Plaque was assessed with each tooth being divided into 6 areas including mesiofacial,facial,distofacial,mesiolingual,lingual,distolingual surfaces.Disclosed plaque was scored for each tooth surface separately as:0 No plaque;1 Slight flecks of plaque at cervical margin of the tooth;2 A thin continuous band of plaque(1 mm or smaller) at cervical margin of tooth;3 A band of plaque wider than 1 mm but covering less than 1/3 of the crown of tooth;4 Plaque covering at least 1/3 but less than 2/3 of crown of tooth;5 Plaque covering 2/3 or more of crown of tooth.Score range 0-5.Lower scores indicate less plaque area.
Time Frame: Baseline to 4 Weeks
Population: ITT (Intent-to-treat) population was the primary analysis population, which included all the participants who were randomized and had at least one post-baseline efficacy evaluation.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Test Product 1: Participants brushed once (1.5g ± 0.05g of toothpaste containing 67 % sodium bicarbonate with 6 herbs plus 923 ppm sodium fluoride), under supervision of study staff for one timed minute.
- Test Product 4: Participants brushed once (1.5g ± 0.05g of toothpaste containing 0% Sodium Bicarbonate without herbs plus 923ppm sodium fluoride), under supervision of study staff for one timed minute.
Arm/Group | Test Product 1 | Test Product 4
Number analyzed (Participants) | 56 | 56
Score on a scale
  Baseline | 2.90 (0.308) | 2.86 (0.309)
  Post Baseline | 1.76 (0.514) | 1.96 (0.470)
  Change from Baseline | -1.13 (0.430) | -0.90 (0.409)
Statistical Analysis 1: Comparison: Test Product 1 vs Test Product 4; Test type: Superiority; p < .0001, ANCOVA — From ANCOVA model with factors for treatment group, period and subject (random effect), and subject-level baseline and period-level baseline; Mean Difference (Net) = -0.21, 95% CI 2-sided [-0.27 to -0.15] — Difference is first named treatment minus second-named treatment such that a negative difference favors the first named treatment

2. Secondary Outcome: Mean Change From Baseline (Pre-brushing to Post Brushing) in Turesky Score After Single Supervised Use for Test Products 1, 2, 3 and 4 After 4 Weeks
Description: The dental examiner used Turesky Modification of the Quigley Hein Index to assess plaque on all gradable teeth.Overall plaque scores were calculated taking average over all tooth sites for participant.Plaque was first disclosed using dye solution followed by disclosing solution.They expectorated and rinsed with 10 mL of water for 10 sec,expectorated again. Plaque was assessed with each tooth being divided into 6 areas including mesiofacial,facial,distofacial,mesiolingual,lingual,distolingual surfaces.Disclosed plaque was scored for each tooth surface separately as:0 No plaque;1 Slight flecks of plaque at cervical margin of the tooth;2 A thin continuous band of plaque(1 mm or smaller) at cervical margin of tooth;3 A band of plaque wider than 1 mm but covering less than 1/3 of the crown of tooth;4 Plaque covering at least 1/3 but less than 2/3 of crown of tooth;5 Plaque covering 2/3 or more of crown of tooth.Score range 0-5.Lower scores indicate less plaque area.
Time Frame: Baseline to 4 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Test Product 1: Participants brushed once (1.5g ± 0.05g of toothpaste containing 67 % sodium bicarbonate with 6 herbs plus 923ppm sodium fluoride), under supervision of study staff for one timed minute.
- Test Product 2: Participants brushed once (1.5g ± 0.05g of toothpaste containing 67% sodium bicarbonate without herbs plus 923ppm sodium fluoride), under supervision of study staff for one timed minute.
- Test Product 3: Participants brushed once (1.5g ± 0.05g of whitening toothpaste containing 62% Sodium Bicarbonate with 6 herbs and 5% w/w silica plus 923ppm Sodium), under supervision of study staff for one timed minute.
Arm/Group | Test Product 1 | Test Product 2 | Test Product 3 | Test Product 4
Number analyzed (Participants) | 56 | 56 | 56 | 56
Score on a scale
  Baseline | 2.90 (0.308) | 2.92 (0.312) | 2.89 (0.304) | 2.86 (0.309)
  Post Baseline | 1.76 (0.514) | 1.78 (0.492) | 1.77 (0.469) | 1.96 (0.470)
  Change from Baseline after 4 weeks | -1.13 (0.430) | -1.14 (0.426) | -1.11 (0.419) | -0.90 (0.409)

ADVERSE EVENTS:
Time Frame: Approximately 15 days (from Screening Visit to 5 days following last visit [Visit 4])
Arm/Group | Test Product 1 | Test Product 2 | Test Product 3 | Test Product 4
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56 | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56 | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 0/56 | 0/56 | 0/56 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.